CLINICAL TRIAL: NCT04992897
Title: Real-world Analysis of Remote Electrical Neuromodulation (REN) for the Acute Treatment of Migraine
Brief Title: Real-world Data Analysis of REN Treatment in Migraine Patients
Status: Completed | Type: Observational
Sponsor: Theranica (Industry)
Collaborators: Georgetown University (Other); Mayo Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: RW002
Record Dates: First submitted 2021-07-04; First posted 2021-08-05 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2021-07

CONDITIONS: Migraine
Keywords: Migraine; headache; REN; Nerivio
MeSH Terms: conditions — Migraine Disorders; Headache

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (4):
- REN-Medication combinations: all evaluable treatments.
  'Treatment' defined as a REN treatment of at least 20 minutes (the nominal duration is 45 minutes).
  'Evaluable treatment' defined as a treatment in which pain levels were reported at baseline and post 2 hours.
  Interventions: Device: Remote Electrical Neuromodulation (REN)
- Consistent efficacy: all users that performed at least 2 evaluable treatments. In order to isolate the effect of REN treatments, this dataset considered only treatments where REN was used as a standalone treatment.
  'Treatment' defined as a REN treatment of at least 20 minutes (the nominal duration is 45 minutes).
  'Evaluable treatment' defined as a treatment in which pain levels were reported at baseline and post 2 hours.
  Interventions: Device: Remote Electrical Neuromodulation (REN)
- Treatment intensity distribution: all treatments.
  'Treatment' defined as a REN treatment of at least 20 minutes (the nominal duration is 45 minutes).
  Interventions: Device: Remote Electrical Neuromodulation (REN)
- Safety: all reported treatment/device-related adverse events (AEs) within the time period.
  Interventions: Device: Remote Electrical Neuromodulation (REN)

INTERVENTIONS:
Device: Remote Electrical Neuromodulation (REN) — Acute migraine treament
  Other Names: Nerivio

SUMMARY:
Data analysis concerning four sets of metrics: A. Per-treatment patterns of REN use as a standalone treatment vs. in combination with medications. B. Per-user Intra-individual consistency of efficacy across multiple treatments (consistency defined as a response to treatment in at least 50% of treatments). C. Distribution of treatment intensity among users (the electroceutical equivalent to treatment dose). D. Prevalence and severity of adverse events.

DETAILED DESCRIPTION:
The REN device The REN device is a wearable device applied to the upper arm and stimulates C and Aδ noxious fibers using a modulated, symmetrical, biphasic, square pulse with a pulse width of 400 μs, modulated frequency of 100-120 Hz, and up to 40 mA output current which can be adjusted by the patient.

Data collection As part of the sign-up process to the Nerivio app, all patients accept the terms of use which specify that providing personal information is done of their own free will, and that their de-identified data may be used for research purposes. Users were not obligated to provide personal information and could treat without providing any feedback. The app includes a secured, personal migraine diary, which enables patients to record and track their migraines and other headaches. At the beginning of each treatment, and again 2 hours after the start of treatment, patients are prompted to record their symptoms, including pain level (none, mild, moderate, severe), functional disability ('No limitation, 'Some limitation', 'Moderate limitation, 'Severe limitation), and indication of which medications, if any, were taken within that 2-hour time window.

Dataset Real-world data of REN treatments collected from patients across the United States who used the REN device.

'Treatment' defined as a REN treatment of at least 20 minutes (the nominal duration is 45 minutes).

'Evaluable treatment' defined as a treatment in which pain levels were reported at baseline and post 2 hours.

Inclusion criteria for each of the different metrics:

A. REN-medication combinations: all evaluable treatments. B. Consistent efficacy: all users that performed at least 2 evaluable treatments. In order to isolate the effect of REN treatments, this dataset considered only treatments where REN was used as a standalone treatment.

C. Intensity stability: all treatments. D. Safety: all reported adverse events (AEs) within the time period.

Outcome measures

Respectively, outcome measures:

A. REN-Medication combinations (prevalence & efficacy):

Medication intake outcomes calculated based on the 2h post-treatment report and comprised of the percentage of treatments in which no rescue medications were used, treatments in which OTC medications were taken, treatments in which triptans were taken, treatments in which other prescription medications were taken, and treatments in which medication intake status was not reported. OTC included acetaminophen, NSAIDs, and combinations of the two, with or without caffeine.

Efficacy outcomes calculated based on the baseline and post-2h reports and comprised of:

(i) consistency of pain relief (decrease in headache from moderate or severe at baseline to mild or no pain); (ii) consistency of pain-freedom (decrease in headache from mild, moderate, or severe at baseline to no pain); (iii) Consistency of improvement in function (improvement in at least one grade between baseline and 2 hours); and (iv) consistency of return to normal function (no functional disability at 2 hours).

B. Consistent efficacy:

Consistency defined as a response of a patient to the treatment in at least 50% of their treated attacks, and calculated for the four efficacy outcomes: (i) consistency of pain relief (ii) consistency of pain-freedom (iii) consistency of improvement in function; and (iv) consistency of return to normal function.

C. Treatment intensity:

The mean intensity of the stimulation collected for all treatments that were 20 minutes or longer, which were performed within the study's time window.

D. Safety:

All adverse events that were reported within the study's period, the following information provided: number of device-related AEs, percentage of the device-related AEs that were mild, moderate, and severe, and percentage of AEs that were serious vs. not serious.

ELIGIBILITY:
Inclusion Criteria:

REN users in the U.S.

Exclusion Criteria:

Cohort 1 REN treatments that were shorter than 20 minutes or did not have a report of pain level.

Cohort 2 Treatments in which medications were taken within 2 hours from REN treatment. Users that had less than 2 REN treatments.

Cohort 3 REN treatments that were shorter than 20 minutes

Cohort 4 All REN sessions, regardless of duration or medication intake.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: REN users across the United States who used Nerivio between October 1st, 2019, and May 24th, 2021.
Sampling Method: Probability Sample
Enrollment: 12151 (Actual)
Dates: Start 2021-06-15 (Actual); Primary Completion 2021-08-07 (Actual); Study Completion 2021-08-10 (Actual)

PRIMARY OUTCOMES:
REN-medication combinations- prevalence | 2 hours from treatment onset
  Medication intake outcomes calculated based on the 2h post-treatment report and comprised of the percentage of treatments in which no rescue medications were used, treatments in which OTC medications were taken, treatments in which triptans were taken, treatments in which other prescription medications were taken, and treatments in which medication intake status was not reported. OTC included acetaminophen, NSAIDs, and combinations of the two, with or without caffeine.
REN-medication combinations- efficacy of the combinations | 2 hours from treatment onset
  The efficacy of treatments in which medications were taken will be calculated based on the 2 hours post-treatment pain report. The overall efficacy rate will be calculated as the percentage of treatments in which response to the treatment was achieved, out of all the treatments.
percentage of users that achieve consistency of efficacy | 2 hours from treatment onset
  Consistency defined as a response of a patient to the treatment in at least 50% of their treated attacks, and calculated for the four efficacy outcomes: (i) consistency of pain relief (ii) consistency of pain-freedom (iii) consistency of improvement in function; and (iv) consistency of return to normal function.
Treatment intensity distribution | 20 minutes from treatment onset
  The mean intensity of the stimulation collected for all treatments that were 20 minutes or longer, which were performed within the study's time window.
Safety (number of users reporting device/treatment-related adverse events) | 20 months
  The percentage of users reporting adverse events, out of the overall number of users, and the severity of the treatment/device-related adverse events.

CONTACTS AND LOCATIONS:
Locations (2):
- Theranica USA Inc, Bridgewater, New Jersey, United States
- Theranica Bio-Electronics, Netanya, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yarnitsky D, Dodick DW, Grosberg BM, Burstein R, Ironi A, Harris D, Lin T, Silberstein SD. Remote Electrical Neuromodulation (REN) Relieves Acute Migraine: A Randomized, Double-Blind, Placebo-Controlled, Multicenter Trial. Headache. 2019 Sep;59(8):1240-1252. doi: 10.1111/head.13551. Epub 2019 May 9. PMID 31074005
- [Background] Tepper SJ, Lin T, Montal T, Ironi A, Dougherty C. Real-world Experience with Remote Electrical Neuromodulation in the Acute Treatment of Migraine. Pain Med. 2020 Dec 25;21(12):3522-3529. doi: 10.1093/pm/pnaa299. PMID 32935848
- [Background] Hershey AD, Lin T, Gruper Y, Harris D, Ironi A, Berk T, Szperka CL, Berenson F. Remote electrical neuromodulation for acute treatment of migraine in adolescents. Headache. 2021 Feb;61(2):310-317. doi: 10.1111/head.14042. Epub 2020 Dec 21. PMID 33349920
- [Background] Nierenburg H, Vieira JR, Lev N, Lin T, Harris D, Vizel M, Ironi A, Lewis B, Wright P. Remote Electrical Neuromodulation for the Acute Treatment of Migraine in Patients with Chronic Migraine: An Open-Label Pilot Study. Pain Ther. 2020 Dec;9(2):531-543. doi: 10.1007/s40122-020-00185-1. Epub 2020 Jul 9. PMID 32648205
- [Background] Rapoport AM, Lin T. Device profile of the Nerivio for acute migraine treatment: overview of its efficacy and safety. Expert Rev Med Devices. 2019 Dec;16(12):1017-1023. doi: 10.1080/17434440.2019.1695599. Epub 2019 Nov 25. PMID 31747304
- [Background] Marmura MJ, Lin T, Harris D, Ironi A, Rosen NL. Incorporating Remote Electrical Neuromodulation (REN) Into Usual Care Reduces Acute Migraine Medication Use: An Open-Label Extension Study. Front Neurol. 2020 Apr 7;11:226. doi: 10.3389/fneur.2020.00226. eCollection 2020. PMID 32318014